CLINICAL TRIAL: NCT03617289
Title: Efficacy of Magnesium Sulfate on Reducing Renal Colic in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Jason Muir, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10080
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-02

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Treatment (Experimental): Receiving Magnesium Sulfate
  Interventions: Drug: Magnesium Sulfate
- Placebo (Placebo Comparator): Receiving Dextrose 5% in Water (D5W)
  Interventions: Drug: D5W

INTERVENTIONS:
Drug: Magnesium Sulfate
  Arms: Treatment
Drug: D5W
  Arms: Placebo

SUMMARY:
To determine if magnesium sulfate paired with an analgesic medication will improve patient pain from renal colic compared with analgesic alone.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old and <100 years old.
* Patients seen in the Emergency Department at Henry Ford Macomb hospital.
* Patients that are A+Ox3.
* Patients who have typical presentation for renal colic.

Exclusion Criteria:

* Age <18 years.
* Patients with a history of dementia, acute delirium or altered mental status.
* Patients with inability to consent to study or inability to fill questionnaire independently.
* Patients with chronic kidney disease and allergies to study drugs.
* Patients that are pregnant (women who are of child-bearing potential will be screened with a urine BHCG).
* Patients with stroke activation or symptoms.
* Patients with trauma activations.
* Patients over the age of 100 years old are excluded as they make up a small percentage of the population and may become identifiable because of their age.
* Imaging study does not show evidence of ureteral stone.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Receiving 15mg ketorolac IV push plus 2g Magnesium Sulfate in 100ml of D5W over 1 hour via pump
- Placebo: Receiving 15mg ketorolac IV push plus dextrose 5% in water (D5W) 100ml over 1 hour via pump
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Receiving Magnesium Sulfate
  Magnesium Sulfate
- Placebo: Receiving D5W
  D5W
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Change
Description: We asked the patient's pain score on a scale of 0-10 with 10 being the highest amount of pain and 0 no pain, before and after treatment (approximately 1 hour). Primary Outcome was the change in score before and after treatment.
Time Frame: 1 hour after the completion of treatment medication (Placebo or Study Drug)
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Treatment: Receiving 15mg ketorolac IV push plus 2g magnesium sulfate in 100ml D5W infused over 1 hour via pump
  Magnesium Sulfate
- Placebo: Receiving 15mg ketorolac IV push plus 100ml D5W infuse over 1 hour via pump
  D5W
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 18 | 19
Units on a Scale | -3.4 (2.7) | -3.6 (3.9)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.771, Wilcoxon (Mann-Whitney) — Threshold for statistical significance set at p<0.05

2. Secondary Outcome: Percentage of Participants Requiring Opiates for Additional Pain Control
Description: We analyzed how many patients required additional pain control with opiates between the two treatment groups.
Time Frame: Any opiate administration required after re-evaluation of pain score after initial treatment with either placebo or study drug
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Receiving 15mg ketorolac IV push plus 100ml D5W infused over 1 hour via pump
  D5W
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 18 | 18
percentage of participants | 16.7 | 47.4
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p < 0.046, Chi-squared — Threshold for statistical significance was set at p<0.05

ADVERSE EVENTS:
Arm/Group | Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No